CLINICAL TRIAL: NCT06490874
Title: Continuous Glucose Monitoring Among Individuals With Gestational Diabetes Treated With Metformin Versus Insulin: Protocol for a Nested Prospective Cohort in the DECIDE RCT (DECIDE CGM)
Brief Title: Continuous Glucose Monitoring (CGM) Substudy of the DECIDE RCT
Acronym: DECIDE CGM
Status: Withdrawn | Type: Observational
Why Stopped: We will focus on parent study
Sponsor: Ohio State University (Other)
Collaborators: The George Washington University Biostatistics Center (Other); DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Kartik K Venkatesh, Associate Professor, Ohio State University
Other Study IDs: 2024H0267
Record Dates: First submitted 2024-06-17; First posted 2024-07-08 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Gestational Diabetes Mellitus; Pregnancy, High Risk
Keywords: Insulin; Pregnancy; Glycemic control; Metformin; Gestational diabetes; Diabetes; Adverse pregnancy outcomes; Continuous glucose monitoring
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- CGM device - Metformin: Individuals will be provided with a CGM device (Dexcom, Inc, San Diego, CA) to be worn for up to 10 days (minimum >5 days) at two pregnancy (randomization to metformin or insulin, late third trimester > 340/7 weeks) and three postpartum timepoints (immediately after delivery, ~6 weeks, and ~2 years). The CGM device will be used in blinded mode for both participants and providers (i.e., neither will be able to see glucose values).
  Interventions: Device: CGM device - Metformin group
- CGM device - Insulin: Individuals will be provided with a CGM device (Dexcom, Inc, San Diego, CA) to be worn for up to 10 days (minimum >5 days) at two pregnancy (randomization to metformin or insulin, late third trimester > 340/7 weeks) and three postpartum timepoints (immediately after delivery, ~6 weeks, and ~2 years). The CGM device will be used in blinded mode for both participants and providers (i.e., neither will be able to see glucose values).
  Interventions: Device: CGM device - Insulin group

INTERVENTIONS:
Device: CGM device - Metformin group — Individuals randomized to metformin will be provided with a CGM device (Dexcom, Inc, San Diego, CA) to be worn for up to 10 days (minimum >5 days) at two pregnancy (randomization to metformin or insulin, late third trimester > 340/7 weeks) and three postpartum timepoints (immediately after delivery, ~6 weeks, and ~2 years).
  Groups: CGM device - Metformin
Device: CGM device - Insulin group — Individuals randomized to insulin will be provided with a CGM device (Dexcom, Inc, San Diego, CA) to be worn for up to 10 days (minimum >5 days) at two pregnancy (randomization to metformin or insulin, late third trimester > 340/7 weeks) and three postpartum timepoints (immediately after delivery, ~6 weeks, and ~2 years).
  Groups: CGM device - Insulin

SUMMARY:
This is a nested multicenter prospective cohort conducted concurrently and in conjunction with the DECIDE two-arm, pragmatic non-inferiority comparative effectiveness Randomized Controlled Trial (RCT) (NCT06445946) of metformin versus insulin among individuals with Gestational diabetes mellitus (GDM) requiring pharmacotherapy for glycemic control. Continuous Glucose Monitoring (CGM)-derived glycemic metric in pregnancy and postpartum will be compared between individuals randomized to metformin versus insulin. In addition, the association between CGM metrics and adverse pregnancy outcomes will be examined. Finally, whether CGM metrics can accurately identify diabetes postpartum compared with an oral glucose tolerance test and hemoglobin A1c will be determined. A total of 300 (150 metformin, 150 insulin) pregnant individuals will be recruited with GDM who require pharmacotherapy to use a blinded CGM device (Dexcom, Inc, San Diego, CA) at two pregnancy (medication randomization, late third trimester) and three postpartum timepoints (delivery, ~6 weeks, and ~2 years).

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is the most frequent metabolic complication of pregnancy, and affects nearly 1 in 10 pregnant individuals in the U.S. annually. GDM increases the risks of both adverse pregnancy and postpartum outcomes for the affected individual and exposed offspring. Following a diagnosis of GDM, individuals are instructed to achieve glycemic control to decrease the risk of adverse pregnancy outcomes through monitoring of blood glucose, dietary modifications, and increased physical activity. However, >1 in 4 individuals with GDM will not achieve targeted glycemic control with diet and behavior changes alone, and require pharmacotherapy.

This is a multicenter prospective observational cohort nested in the DECIDE randomized controlled trial (NCT06445946). DECIDE is a two-arm, pragmatic non-inferiority comparative effectiveness RCT of metformin versus insulin to prevent adverse pregnancy outcomes and to confirm postpartum safety among individuals with GDM who require pharmacotherapy to achieve glycemic control. This trial will determine whether metformin is not inferior to insulin in reducing adverse pregnancy outcomes and is comparably safe for exposed pregnant individuals and their children. This substudy will be conducted concurrently and in conjunction with the parent study. A subset of 300 individuals (150 metformin, 150 insulin) will be enrolled in this substudy from the 1,572 individuals from the parent trial.

Primary aim:

To compare CGM-derived glycemic profiles (primary outcome: time in range of 63 to 140 mg/dL; secondary outcomes (mean glucose, coefficient of variation, and percentage of time below the target glucose range or above the target glucose range) in pregnancy between individuals with GDM randomized to metformin versus insulin.

Secondary aims:

To examine the association between CGM metrics and adverse pregnancy outcomes (large-for-gestational-age at birth, neonatal hypoglycemia, and hyperbilirubinemia, hypertensive disorder of pregnancy, preterm birth <37 weeks, NICU admission, neonatal mechanical ventilation, neonatal oxygen support, neonatal respiratory distress syndrome).

To examine whether CGM metrics can identify diabetes and postpartum cardiometabolic outcomes (prediabetes, type 2 diabetes, impaired glucose tolerance, impaired fasting glucose, hypertension, obesity, and cholesterol abnormalities) compared with an oral glucose tolerance test or hemoglobin A1c.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation. Twin reduction to singleton, either spontaneously or therapeutically, is eligible if it occurred before 14 weeks gestational age.
* Age >18 years
* Gestational age at randomization between 200/7 - 316/7 weeks based on project gestational age.
* GDM diagnosis between 200/7 - 316/7 weeks based on project gestational age.
* Requires medication for glucose control defined as ≥30% elevated glucose values (either fasting or postprandial or both) in the week prior to randomization per determination of the provider or documented in the medical record.
* Patient willingness and ability to attend 2-year follow-up visit.
* Patient willingness to wear and return a blinded CGM device. It is possible that some enrolled individuals may choose to use a separate CGM device for glucose monitoring as part of clinical care.

Exclusion Criteria:

* Renal disease (serum creatinine >1.3 mg/dL) due to the potential impact of metformin on renal function.
* Major structural malformation of the fetus.
* Known fetal aneuploidy based on invasive testing or positive for aneuploidy on cell-free fetal DNA screening.
* Contraindication to metformin or insulin, including: history of lactic acidosis, intractable nausea and vomiting, prior documented allergy and/or anaphylaxis.
* Pregestational diabetes documented in the medical record, GDM diagnosis <20 weeks, or prior A1c>6.5%
* Fasting hyperglycemia >115 mg/dl for ≥50% of fasting glucose values in the past week (due to the high risk of metformin failure with fasting hyperglycemia).
* Enrolled in a trial that influences primary study outcomes of the parent DECIDE trial (composite neonatal outcome at delivery or childhood body mass index at 2 years).
* Prenatal care or delivery planned at a location where access to the complete electronic medical record will not be available to research staff.
* Language barrier (appropriate translation resources unavailable at the site).
* Participation in this trial in a previous pregnancy. Patients who were screened in a previous pregnancy, but not randomized, may be included.
* In addition, individuals who report a prior allergy or sensitivity to CGM will also be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is restricted to pregnant individuals with GDM.
Study Population: A subset of 300 individuals (150 metformin, 150 insulin) will be consecutively enrolled in participating sites to this substudy from the 1,572 individuals from the parent DECIDE trial (NCT06445946).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Time in range (TIR) | From medication randomization till late third trimester, up to 14 weeks
  Percent of time CGM readings are within the pregnancy target glucose range of 63 to 140 mg/dL. This outcome will be assessed as a continuous measure in increments of 1%.

SECONDARY OUTCOMES:
Coefficient of variation (CV) | From medication randomization till 2 years postpartum, up to 40 months.
  Percent of glycemic variability calculated as the standard deviation (SD) of glucose values divided by the mean glucose in the same observation period, continuous measure
Time below range (TBR) | From medication randomization till 2 years postpartum, up to 40 months.
  Percent of CGM readings and time below the target glucose range of <63 mg/dL, continuous measure
Time above range (TAR) | From medication randomization till 2 years postpartum, up to 40 months.
  Percent of CGM readings and time above the target glucose range of >140 mg/dL, continuous measure
Large-for-gestational-age at birth | At delivery
  LGA will be defined as a birthweight ≥90th%tile for gestational age based on a US birth certificate reference adjusted for parity and/or fetal sex.
Hypoglycemia | <24 hours after birth
  Neonatal hypoglycemia will be defined as a blood glucose <35 mg/dL or treatment <24 hours after birth with either IV, PO, or gel glucose therapy.
Hyperbilirubinemia | Within one week after birth
  Neonatal hyperbilirubinemia will be defined as treated with phototherapy or exchange transfusion in the first postnatal week and either treatment in the first postnatal week or kernicterus.
Hypertensive disorder of pregnancy | Randomization to delivery
  HDP will include either gestational hypertension or preeclampsia. Gestational hypertension will be defined as: systolic blood pressure of 140 mm Hg or more or diastolic blood pressure of 90 mm Hg or more on two occasions at least 4 hours apart after 20 weeks of gestation in a woman with a previously normal blood pressure. Preeclampsia will be defined as: above blood pressure criteria AND proteinuria (300 mg or more per 24 hour urine collection, protein/creatinine ratio of 0.3 mg/dL or more, or dipstick reading of 2+) OR thrombocytopenia (platelet count less than 100 109/L), renal insufficiency (serum creatinine greater than 1.1 mg/dL or a doubling of the serum creatinine concentration in the absence of other renal disease), impaired liver function (elevated blood concentrations of liver transaminases to twice normal concentration), pulmonary edema, new-onset headache or visual symptoms not attributed to other diagnoses.
Preterm birth | At birth
  Preterm birth <37 weeks and <34 weeks based on project gestational age.
Requiring mechanical ventilation | <72 hours after birth
  Intubation, continuous positive airway pressure (CPAP) or high-flow nasal cannula (HFNC) for ventilation or cardiopulmonary resuscitation within first 72 hours of birth.
NICU admission | Birth to infant date of delivery discharge (length of NICU admission will vary for each infant )
  Admitted to NICU or intermediate nursery ≥72 hours, any indication.
Oxygen support | <72 hours after birth
  Requiring oxygen support.
Respiratory distress syndrome | Anytime during the first 72 hours after birth
  Signs of respiratory distress with oxygen requirement and confirmed by chest x-ray.
Treatment supplementation | From randomization to delivery
  Insulin use among individuals randomized to metformin between randomization and delivery.
Type 2 diabetes (T2D) | From delivery to 2 years postpartum
  A1c > 6.5% OR fasting plasma glucose > 126 mg/dL OR OGTT > 200 mg/dL OR prior diagnosis per patient report.
Prediabetes | From delivery to 2 years postpartum
  A1c 5.7% to 6.4% OR fasting plasma glucose 100 mg/dl to 125 mg/dL OR OGTT 140 to 199 mg/dL.
Impaired glucose tolerance (IGT) | From delivery to 2 years postpartum
  OGTT 2-hour value of 140 to 199 mg/dL32
Impaired fasting glucose (IFG) | From delivery to 2 years postpartum.
  OGTT value of 100 to 125 mg/dL.
Obesity overall and by class | 2 years postpartum
  Weight and height will be combined to report BMI in kg/m^2. BMI per the following classifications will be assessed: Normal or underweight: < 25 kg/m2; Overweight: 25 to < 30 kg/m2; Class 1: 30 to < 35 kg/m2; Class 2: 35 to < 40 kg/m2; and Class 3: 40 kg/m2 or greater.
Hypertension | 2 years postpartum
  Per American Heart Association criteria as below and/or antihypertensive medication or prior diagnosis per patient report, and defined as: Elevated: Systolic between 120-129 and diastolic less than 80 mm Hg; Stage 1: Systolic between 130-139 or diastolic between 80-89 mm Hg; and Stage 2: Systolic at least 140 or diastolic at least 90 mm Hg.
Cholesterol | 2 years postpartum
  Fasting state, defined as a continuous measure and dichotomous at the following thresholds for each component: Total cholesterol: > 200 mg/dL; LDL cholesterol: > mg/dL; HDL cholesterol: < 40 mg/dL; Triglycerides: > 200 mg/dL.
Mean glucose | From medication randomization till 2 years postpartum, up to 40 months.
  Mean glucose in mg/dL per CGM readings, continuous measure

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Venkatesh, MD, PhD, Principal Investigator — Ohio State University; Donna Gregory, RNC, BSN, Study Director — Ohio State University
Locations (4):
- United States (4):
  - University of Alabama, Tuscaloosa, Alabama
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio
  - Premier Health - Miami Valley Hospital, Dayton, Ohio

IPD SHARING:
Plan to Share IPD: No